CLINICAL TRIAL: NCT03606837
Title: Exploratory, Single-institution Study, Comparing 68Ga-RM2 PET/CT Versus 68Ga-PSMA-617 PET/CT in Patients Diagnosed With Intermediate Risk Prostate Cancer Candidates for Radical Prostatectomy
Brief Title: 68Ga-RM2 Compared to 68Ga-PSMA-617 PET/CT for Intermediate Risk Prostate Cancer Imaging
Acronym: PROSTATEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX2016/46
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; 68Ga-RM2; 68Ga-Prostate Specific Membrane Antigen; PET/CT; Prostate cancer imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/CT Imaging (Experimental)
  Interventions: Drug: 68Ga-PSMA-617 PET/CT; Drug: 68Ga-RM2 PET/CT

INTERVENTIONS:
Drug: 68Ga-PSMA-617 PET/CT — PET/CT Imaging with 68Ga-PSMA-617 injection
Drug: 68Ga-RM2 PET/CT — PET/CT Imaging with 68Ga-RM2 injection

SUMMARY:
Patients with primary intermediate risk prostate cancer for whom radical prostatectomy is indicated, will be invited to participate to the present study.

Positron Emission Tomography coupled with scanner (PET-CT) using a radiotracer : 68Ga-RM2 and Positron Emission Tomography coupled with scanner (PET-CT) using another radiotracer : 68Ga-PSMA-617, will be scheduled.

DETAILED DESCRIPTION:
European Association of Urology (EAU) Guidelines for initial staging of intermediate risk prostate cancer (Gleason score 3+4 and 4+3) include tomodensitometry (CT scan), magnetic resonance imaging (MRI) and bone scintigraphy. However, this group of tumor is highly heterogeneous. A distinction exist between tumors with Gleason score 3+4 (lower risk) and 4+3 which may be closer to high risk prostate cancer.

Consequently, management of these two sub-groups of tumors differs. The key point for optimal management of these tumors is to get specific and non-invasive molecular tools for better classification and stratification. This is of critical importance for personalized treatment decision-making.

Novel innovative radiotracers are today available for prostate cancer imaging notably small molecules, radiolabeled with 68Ga, targeting the prostate specific membrane antigen (PSMA) or antagonists, radiolabeled with 68Ga, targeting the Gastrin-Releasing Peptide receptor (GRP-R, a bombesin receptor subtype).

There are on growing evidences that Positron Emission Tomography coupled to Computed Tomography (PET-CT) with radiolabeled prostate specific membrane antigen analogues (PSMA) could be more sensitive and more specific for the detection of lymph node metastasis in high-risk cancers, as shown with PSMA-617 in recent studies.

ELIGIBILITY:
Inclusion criteria:

15 patients divided in :

* 7 patients with favourable intermediate risk prostate cancer (cT2b or Gleason score 7 (3+4) or PSA value 10-20 ng/mL, Briganti 5-20%,)
* 8 patients with unfavourable intermediate risk prostate cancer (cT2b or Gleason score 7 (4+3) or PSA value 10-20 ng/mL, Briganti 5-20%,)
* who are candidate for radical prostatectomy after discussion in multidisciplinary committee
* covered by the national health insurance system
* with freely written informed consent obtained

Exclusion criteria:

* Any kind of previous treatment for prostate cancer (hormonal treatment, EBRT, brachytherapy, cryotherapy, etc…);
* Patient with prostate cancer not candidate for radical prostatectomy and/or unable to benefit from surgery
* Freedom privated patient
* Patient under legal protection or unable to express its own consent
* Known contraindication to radiopharmaceuticals and / or excipients ……

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Median Standardized Uptake Value (SUV) | Day 0 (inclusion) or Day 2 to 21 (Visit 2)
  Uptake intensity of 68Ga-PSMA-617

SECONDARY OUTCOMES:
Gleason score | Day 3 to 60 (Last visit)
Receptor density Bmax | Day 0 (inclusion) or Day 2 to 21 (Visit 2)
Local radioactive concentration (cpm) | Day 0 (inclusion) or Day 2 to 21 (Visit 2)
Immunoreactive score (IRS) | Day 3 to 60 (Last visit)
New World Health Organization 2016 classification | Day 3 to 60 (Last visit)

CONTACTS AND LOCATIONS:
Overall Officials: Henri CLERMONT-GALLERANDE, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No